CLINICAL TRIAL: NCT01382238
Title: Relative Bioavailability Study of a Tablet Formulation vs. Pediatric Granule Formulation of Dolutegravir 50 mg and Effect of Different Types of Water Plus Infant Formula on the Pediatric Granule Formulation in Healthy Male and Female Volunteers
Brief Title: Relative Bioavailability Study of a Pediatric Granule Formulation of Dolutegravir
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Collaborators: Shionogi (Industry); GlaxoSmithKline (Industry)
Responsible Party: Cheri Hudson; Clinical Disclosure Advisor, GSK Clinical Disclosure
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 114556; NCT01371500 (obsolete NCT alias)
Record Dates: First submitted 2011-06-23; First posted 2011-06-27 (Estimated); Last update posted 2011-09-19 (Estimated); Status verified 2011-09

CONDITIONS: Infections, Human Immunodeficiency Virus and Herpesviridae
Keywords: dolutegravir; pediatric; granule formulation; GSK1349572; HIV
MeSH Terms: conditions — Infections; Acquired Immunodeficiency Syndrome | interventions — dolutegravir; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single arm (Experimental): Subjects will have a screening visit within 30 days prior to the first dose of study drug, five treatment periods containing a single dose of study drug, followed by 48 hours of serial PK collection. In the 5 treatment periods subjects will receive DTG granule formulation 1) directly to mouth; 2) with purified water; 3) with Contrex brand water; and 4) with milk-based infant formula. They will also receive the current 50 mg tablet formulation administered with tap water. These treatments will be administered in a random order. Subjects will check out of the unit on Day 3 after the 48 hour PK sample in each period. Study periods will be separated by at least 5 days. Subjects will have a follow-up visit 5-7 days after last dose of DTG given.
  Interventions: Drug: Dolutegravir 50 mg tablet; Drug: Dolutegravir 50 mg oral granules

INTERVENTIONS:
Drug: Dolutegravir 50 mg tablet — Dolutegravir is an experimental drug in the integrase inhibitor class for the treatment of HIV.
Drug: Dolutegravir 50 mg oral granules — Dolutegravir is an experimental drug in the integrase inhibitor class for the treatment of HIV.

SUMMARY:
Dolutegravir (DTG, GSK1349572) is an integrase inhibitor currently in Phase 3 clinical trials for the treatment of human immunodeficiency virus (HIV) infection. A granule formulation has been developed as an alternative to the current tablet formulation for administration in pediatric populations.

This is a single-center, randomized, open-label, 5-way crossover study in healthy adult subjects. The study will evaluate the relative bioavailability of a 50 mg granule formulation of dolutegravir when administered 1) directly to mouth; 2) with purified water; 3) with Contrex brand water; and 4) with milk-based infant formula compared to the current 50 mg tablet formulation administered with tap water. Safety evaluations and serial PK samples will be collected during each treatment period. A taste assessment of the granule will also be performed. A follow-up visit will occur 5-7 days after the last dose of study drug.

Pharmacokinetic assessments during the study will include area under the concentration-time curve from time zero (pre-dose) extrapolated to infinite time (AUC(0-infinity)), area under the concentration-time curve from time zero (pre-dose) to last time of quantifiable concentration within a subject across all treatments (AUC(0-t)), maximum observed concentration (Cmax), terminal phase half-life (t½), lag time before observation of drug concentrations in sampled matrix (tlag), time of occurrence of Cmax (tmax), concentration at 24 hours post-dose (C24), and apparent clearance following oral dosing (CL/F).

DETAILED DESCRIPTION:
ViiV Healthcare is the new sponsor of this study, and GlaxoSmithKline is in the process of updating systems to reflect the change in sponsorship

ELIGIBILITY:
Inclusion Criteria:

* ALT, alkaline phosphatase and bilirubin less than or equal to 1.5x upper limit of normal (ULN) (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%). A single repeat is allowed for eligibility determination.
* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring.
* Male or female between 18 and 65 years of age inclusive, at the time of signing the informed consent.
* A female subject is eligible to participate if she is of: Non-childbearing potential or child-bearing potential and agrees to use an appropriate contraception method for an appropriate period of time (as determined by the product label or investigator) prior to the start of dosing to sufficiently minimize the risk of pregnancy at that point. Female subjects must agree to use contraception until the follow-up visit.
* Body weight greater than or equal to 50 kg for males and 45 kg for females and body mass index (BMI) within the range 18.5- 31.0 kg/m2 (inclusive).
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.

Exclusion Criteria:

* The subject has a positive pre-study drug/alcohol screen. A minimum list of drugs that will be screened for include amphetamines, barbiturates, cocaine, opiates, cannabinoids and benzodiazepines.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* History of sensitivity to any of the study medications, or components thereof, or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* If heparin is used during PK sampling, subjects with a history of sensitivity to heparin or heparin-induced thrombocytopenia should not be enrolled.
* History of regular alcohol consumption within 6 months of the study defined as an average weekly intake of >14 drinks/week for men or >7 drinks/week for women. - Consumption of red wine, seville oranges, grapefruit or grapefruit juice from 7 days prior to the first dose of study medication.
* Pregnant females as determined by positive serum or urine human chorionic gonadotrophin (hCG) test at screening or prior to dosing.
* Lactating females.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* Subjects with a pre-existing condition interfering with normal gastrointestinal anatomy or motility, hepatic and/or renal function, that could interfere with the absorption, metabolism, and/or excretion of the study drugs. Subjects with a history of cholecystectomy, peptic ulceration, inflammatory bowel disease or pancreatitis should be excluded.
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening.
* A positive test for HIV antibody.
* History of Gilbert's disease.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* The subject's systolic blood pressure is outside the range of 90-140mmHg, or diastolic blood pressure is outside the range of 45-90mmHg or heart rate is outside the range of 50-100bpm for female subjects or 45-100 bpm for male subjects. A single repeat is allowed for eligibility determination.
* Exclusion criteria for screening ECG within protocol limits.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-06; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Plasma DTG AUC(0-infinity), AUC(0-t), and Cmax | 48 hours post dose

SECONDARY OUTCOMES:
Plasma DTG t½, tlag, tmax, C24, and CL/F | 48 hours post dose
Safety and tolerability parameters as assessed by change from baseline in 12-lead ECG and vital signs (BP and HR), number of subjects with adverse events and toxicity grading of clinical laboratory tests | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (1):
- GSK Investigational Site, Austin, Texas, United States